CLINICAL TRIAL: NCT03894215
Title: A Two-arm, Randomized, Non-comparative, Phase 2 Trial of AGEN2034 (Anti-PD-1) as a Monotherapy or Combination Therapy With AGEN1884 (Anti- CTLA4) or With Placebo in Women With Recurrent Cervical Cancer (Second Line) - RaPiDS
Brief Title: RaPiDS- A Phase 2 Study of Anti-PD-1 Independently or in Combination With Anti-CTLA-4 in Second-Line Cervical Cancer
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Agenus Inc. (Industry)
Collaborators: GOG Foundation (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: C-750-01/GOG-3028
Expanded Access: NCT05572970 (Available)
Record Dates: First submitted 2019-03-19; First posted 2019-03-28 (Actual); Last update posted 2025-02-20 (Actual); Status verified 2025-02

CONDITIONS: Cervical Cancer
MeSH Terms: conditions — Uterine Cervical Neoplasms | interventions — balstilimab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- AGEN2034 + Placebo (Experimental): AGEN2034 administered with placebo monotherapy: approximately 100 patients.
  Interventions: Drug: AGEN2034
- AGEN2034 + AGEN1884 (Experimental): AGEN2034 administered in combination with AGEN1884 (combination therapy): approximately 100 patients.
  Interventions: Drug: AGEN2034; Drug: AGEN1884

INTERVENTIONS:
Drug: AGEN2034 — PD-1 antibody
Drug: AGEN1884 — CTLA-4 antibody
  Arms: AGEN2034 + AGEN1884

SUMMARY:
This is a randomized, blinded, non-comparative, two-arm Phase 2 clinical trial to assess the efficacy and safety of AGEN2034 administered with placebo (Treatment Arm 1 - monotherapy) or with AGEN1884 (Treatment Arm 2- combination therapy) for treatment of patients with advanced cervical cancer who relapsed or progressed after receiving first-line platinum-based chemotherapy. The study is not intended to compare the efficacy of the 2 experimental arms. Rather, the efficacy of each arm will be evaluated against its relevant historical controls as appropriate.

DETAILED DESCRIPTION:
This is a randomized, blinded, non-comparative, two-arm Phase 2 clinical trial to assess the efficacy and safety of AGEN2034 administered with placebo (Treatment Arm 1 - monotherapy) or with AGEN1884 (Treatment Arm 2- combination therapy) for treatment of patients with advanced cervical cancer who relapsed or progressed after receiving first-line platinum-based chemotherapy. The study is not intended to compare the efficacy of the 2 experimental arms. Rather, the efficacy of each arm will be evaluated against its relevant historical controls as appropriate Patients will receive AGEN2034 with placebo as a monotherapy or with AGEN1884 as combination therapy for a maximum of 24 months or until confirmed progression, unacceptable toxicity, or any criterion for stopping the study drug or withdrawal from the trial occurs. Placebo administration in Treatment Arm 1 (AGEN 2034 monotherapy) of the study is intended to preserve the integrity of the investigators' interpretation of the efficacy and safety data by eliminating biases in disease assessment monitoring, declaration of disease progression, and assessment of toxicities. Therefore, it is understood that investigators, patients, and research personnel will not know whether patients have received AGEN2034/placebo (Treatment Arm 1) or AGEN2034/AGEN1884 (Treatment Arm 2).

An Independent Data Monitoring Committee (IDMC) will evaluate safety and efficacy. An IRRC will be established to adjudicate tumor response.

ELIGIBILITY:
Inclusion Criteria:

1. Voluntarily agree to participate by giving written informed consent. (Participation in pharmacogenomics testing is optional).
2. Be ≥18 years of age.
3. Diagnosis:

   1. Have (1) a histologically or cytologically confirmed diagnosis of squamous-cell carcinoma, adenosquamous carcinoma, or adenocarcinoma of the cervix, and (2) metastatic, locally advanced, and/or unresectable disease at the time of enrollment. Histologic confirmation of the original primary tumor is required via pathology report.

      Note: The following cervical tumors are not eligible: minimal deviation/adenoma malignum, gastric type adenocarcinoma, clear cell carcinoma, and mesonephric carcinoma.
   2. Has cervical cancer and has relapsed after a platinum- based treatment (first line) regimen for advanced (recurrent, unresectable, or metastatic) disease.
4. Measurable Disease:

   a. Have measurable disease on imaging based on RECIST version 1.1 by Investigator assessments and independent central radiologic review.

   Note: Patients without centrally confirmed measurable disease at baseline will not be eligible for this trial.

   Note: Patients must have at least 1 "target lesion" to be used to assess response, as defined by RECIST version 1.1. Tumors within a previously irradiated field will be designated as "non-target" lesions unless progression is documented, or a biopsy is obtained to confirm persistence at least 90 days following completion of radiation therapy.
5. Have a life expectancy of at least 3 months and an Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
6. Have adequate organ function as indicated by the following laboratory values:

   1. Adequate hematological function defined by absolute neutrophil count (ANC) > 1.5 x 10^9/L, platelet count > 100 x 10^9/L, and hemoglobin >8 g/dL (without transfusions within 1 week of first dose).
   2. Adequate hepatic function based by a total bilirubin level ≤ 1.5 the institutional upper limit of normal (IULN), aspartate aminotransferase (AST) level ≤ 2.5 x IULN, alanine aminotransferase (ALT) level ≤ 2.5 x IULN, and alkaline phosphatase ≤ 2.5 IULN and albumin ≥3.0 mg/dL.
   3. Adequate renal function defined as creatinine ≤ 1.5 × upper limit of normal (ULN) OR measured or calculated creatinine clearance ≥ 40 mL/minute per Institutional standard. Assessment methods should be recorded.
   4. Adequate coagulation defined by international normalized ratio (INR) or prothrombin time ≤ 1.5 x IULN (unless the patient is receiving anticoagulant therapy); and activated partial thromboplastin time (aPTT) ≤ 1.5 x IULN (unless the patient is receiving anticoagulant therapy)
7. Has no history of another primary malignancy, with the exception of:

   1. Malignancy treated with curative intent and with no known active disease ≥ 3 years before the first dose of study drug and of low potential risk for recurrence.
   2. Adequately treated non-melanoma skin cancer or lentigo maligna without evidence of disease and superficial bladder cancer.
8. Patients must provide a sufficient and adequate FFPE tumor tissue sample preferably from the most recent biopsy of a tumor lesion, collected either at the time of or after the diagnosis of advanced or metastatic disease has been made AND from a site not previously irradiated. Archival tumor tissue must be ≤ 3 years old. If no tumor tissue is available, a fresh biopsy will be required (See Section 7.2.3.1 for details).

   Note: Tissue from core biopsy or excisional biopsy or from resection is required.
9. Patients must have a negative serum pregnancy test at screening (within 72 hours of first dose of study medication) if of childbearing potential or be of non-childbearing potential. Non-childbearing potential is defined as (by other than medical reasons):

   1. ≥45 years of age and has not had menses for greater than 1 year,
   2. Amenorrheic ≥ 2 years without a hysterectomy and oophorectomy and a follicle-stimulating hormone (FSH) value in the postmenopausal range upon pretrial (screening) evaluation,
   3. History of hysterectomy, oophorectomy or tubal ligation.
   4. Definitive pelvic radiation for the treatment of cervical cancer.
10. If of childbearing potential, female patients must be willing to use 2 adequate barrier methods throughout the study, starting with the screening visit through 120 days after the last dose of study treatment. Note: Abstinence is acceptable if this is the established and preferred contraception for the patient.
11. Is willing and able to comply with the requirements of the protocol.

Exclusion Criteria:

The patient must be excluded from participating in the trial if the patient:

1. Is currently participating and receiving study therapy or has participated in a study of an investigational agent and received study therapy or used an investigation device within 4 weeks of the first dose of treatment.
2. Has an inadequate washout period prior to first dose of study drug defined as:

   1. Received systemic cytotoxic chemotherapy or biological therapy within 3 weeks before first dose,
   2. Received radiation therapy within 3 weeks before first dose, or
   3. Had major surgery within 4 weeks before first dose.
3. Has received prior therapy with:

   1. Any antibody/drug targeting T-cell co-regulatory proteins (immune checkpoints) such as anti-PD-1, anti-PD-L1, or anti- cytotoxic T-lymphocyte antigen 4 (CTLA-4) antibodies
   2. More than 1 systemic treatment regimen for the advanced (recurrent, unresectable, or metastatic) cervical cancer for which the patient is considered for the study.
4. Has persisting toxicity related to prior therapy of National Cancer Institute Common Terminology Criteria for Adverse Events version 5.0 (NCI-CTCAE) Grade >1 severity.

   Note: Sensory neuropathy or alopecia of Grade ≤2 is acceptable.
5. Is expected to require any other form of systemic or localized antineoplastic therapy while on trial (including maintenance therapy with another agent, radiation therapy, and/or surgical resection).
6. Has known severe hypersensitivity reactions to fully human monoclonal antibodies (NCI-CTCAE Grade ≥3), any history of anaphylaxis, or uncontrolled asthma.
7. Has received systemic corticosteroid therapy ≤ 7 days prior to the first dose of trial treatment or receiving any other form of systemic immunosuppressive medication (corticosteroid use on study for management of immune-related adverse events (AE), and/or a premedication for IV contrast allergies/reactions is allowed). Patients who are receiving daily corticosteroid replacement therapy are an exception to this rule. Daily prednisone at doses of up to 5 mg or equivalent hydrocortisone dose are examples of permitted replacement therapy.
8. Has a central nervous system (CNS) tumor, metastasis(es), and/or carcinomatous meningitis identified either on the baseline brain imaging obtained during the screening period OR identified prior to consent.

   Note: Patients with history of brain metastases that have been treated may participate provided they show evidence of stable supra-tentorial lesions at screening (based on 2 sets of brain images, performed ≥ 4 weeks apart, and obtained after the brain metastases treatment). In addition, any neurologic symptoms that developed either as a result of the brain metastases or their treatment must have resolved or be minimal and be expected as sequelae from treated lesions. For individuals who received steroids as part of brain metastases treatment, steroids must be discontinued ≥ 7 days prior to first dose of study drug.
9. Has active or history of autoimmune disease that has required immunosuppressive systemic treatment within 2 years of the start of trial treatment (i.e. with use of disease modifying agents, corticosteroids or immunosuppressive drugs). Replacement therapy (i.e., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of immunosuppressive systemic treatment.

   Note: Patients with diabetes type 1, vitiligo, psoriasis, hypo-, or hyperthyroid disease not requiring immunosuppressive treatment are eligible.
10. Has had an allogeneic tissue/solid organ transplant.
11. Has or had interstitial lung disease (ILD) OR has had a history of pneumonitis that has required oral or IV corticosteroids.
12. Has an active infection requiring intravenous (IV) systemic therapy.
13. Has known history of Human Immunodeficiency Virus (HIV) (HIV 1/2 antibodies).
14. Has known active Hepatitis B (HBV), Hepatitis C (HCV), or tuberculosis. Active Hepatitis B is defined as a known positive HBsAg result. Active Hepatitis C is defined by a known positive Hep C Ab result and known quantitative HCV ribonucleic acid (RNA) results greater than the lower limits of detection of the assay.
15. Has clinically significant (i.e., active) cardiovascular disease: cerebral vascular accident/stroke or myocardial infarction within 6 months of enrollment, unstable angina, congestive heart failure (New York Heart Association class ≥II), or serious uncontrolled cardiac arrhythmia requiring medication.
16. Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the trial, interfere with the patient's participation for the full duration of the trial, or is not in the best interest of the patient to participate, in the opinion of the treating investigator.
17. Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.
18. Is, at the time of signing informed consent, a regular user (including "recreational use") of any illicit drugs or had a recent history (within the last year) of substance abuse (including alcohol). Medicinal marijuana use is not considered "illicit" and is allowed to be utilized prior to and during enrollment.
19. Is legally incapacitated or has limited legal capacity.
20. Is pregnant or breastfeeding or expecting to conceive within the projected duration of the trial, starting with the screening visit through 120 days after the last dose of the study drug.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Only female
Enrollment: 212 (Estimated)
Dates: Start 2019-06-01 (Actual); Primary Completion 2025-08 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate | 48 months
  To assess the Objective Response Rate (ORR) to the treatment of AGEN2034 (anti-PD-1) administered with placebo (Treatment Arm 1 - monotherapy), or with AGEN1884 (anti-CTLA4) (Treatment Arm 2 - combination therapy), defined as the binomial proportion of intent to treat (ITT) patients with best overall response (BOR) of complete response (CR) or partial response (PR), in women with recurrent/persistent/metastatic cervical cancer who have progressed following first-line therapy. BOR will be determined by the Independent Radiology Review Committee (IRRC), according to Response Evaluation Criteria in Solid Tumors version 1.1 (RECIST 1.1).

SECONDARY OUTCOMES:
Frequency, severity and duration of treatment-emergent AEs | 48 months
  To confirm the safety and tolerability of AGEN2034 administered with placebo (Treatment Arm 1 - monotherapy) or with AGEN1884 (Treatment Arm 2 - combination therapy) in patients with recurrent, progressive second-line cervical cancer.
DOR per RECIST 1.1 | 48 months
  To assess duration of response (DOR), stable disease (SD), duration of stable disease and disease control rate (DCR), overall survival (OS), and progression-free survival (PFS) per RECIST 1.1 for AGEN2034 administered with placebo (Treatment Arm 1 - monotherapy) or with AGEN1884 (Treatment Arm 2 - combination therapy).
Time to Confirmed Progression | 48 months
  To estimate the time to confirmed progression by the investigator per iRECIST for AGEN2034 administered with placebo (Treatment Arm 1 - monotherapy) or with AGEN1884 (Treatment Arm 2 - combination therapy).
Immunogenicity of AGEN2034 | 48 months
  To evaluate the immunogenicity of AGEN2034 administered with placebo (Treatment Arm 1 - monotherapy) or with AGEN1884 (Treatment Arm 2 - combination therapy) and to correlate it to exposure and biological activity.
Maximum observed drug concentration at steady state (Cmax-ss) | 48 months
  To characterize AGEN2034 and AGEN1884 pharmacokinetics (PK).
Minimum observed drug concentration at steady-state (Cmin-ss) | 48 months
  To characterize AGEN2034 and AGEN1884 pharmacokinetics (PK).
Area under the concentration-time curve within time span t1 to t2 at steady-state (AUC(τ1-τ2)-ss) | 48 months
  To characterize AGEN2034 and AGEN1884 pharmacokinetics (PK).
Area under the drug concentration-time curve from time zero to time t (AUC(0-t)) | 48 months
  To characterize AGEN2034 and AGEN1884 pharmacokinetics (PK).
Area under the drug concentration-time curve from time zero to infinity (AUC(0-∞)) | 48 months
  To characterize AGEN2034 and AGEN1884 pharmacokinetics (PK).
Time to maximum drug concentration (tmax) | 48 months
  To characterize AGEN2034 and AGEN1884 pharmacokinetics (PK).
Terminal disposition rate constant (λz) | 48 months
  To characterize AGEN2034 and AGEN1884 pharmacokinetics (PK).
Terminal elimination half-life (t1/2) | 48 months
  To characterize AGEN2034 and AGEN1884 pharmacokinetics (PK).
Systemic clearance (CL) | 48 months
  To characterize AGEN2034 and AGEN1884 pharmacokinetics (PK).
Volume of distribution (Vd) | 48 months
  To characterize AGEN2034 and AGEN1884 pharmacokinetics (PK).
Quality of Life Assessment per FACT-Cx | 35 months
  To assess quality of life in the treated population using the Functional Assessment of Cancer Therapy - Cervical Cancer Trial Outcome Index (FACT-Cx)
Quality of Life Assessment per BPI | 35 months
  To assess quality of life in the treated population using Brief Pain Inventory (BPI)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Agenus Inc.
Locations (68):
- United States (42):
  - University of Alabama at Birmingham School of Medicine, Birmingham, Alabama
  - University of South Alabama Mitchell Cancer Institute, Mobile, Alabama
  - Arizona Oncology - Biltmore Cancer Center, Phoenix, Arizona
  - Arizona Oncology - Tucson - Wilmot Road Location, Tucson, Arizona
  - University of California, San Diego (UCSD) - Moores Cancer Center, La Jolla, California
  - UCLA- Women's Health Clinical Research Unit (WHCRU), Los Angeles, California
  - Gynecologic Oncology Associates, Newport, California
  - California Pacific Medical Center, San Francisco, California
  - University of California, San Francisco Medical Center, San Francisco, California
  - Baptist MD Anderson Cancer Center, Jacksonville, Florida
  - Moffitt Cancer Center, Tampa, Florida
  - Northside Hospital, Atlanta, Georgia
  - St Joseph's Hospital, Savannah, Georgia
  - Community Health Network - North Cancer Center, Indianapolis, Indiana
  - University of Kentucky Albert B. Chandler Hospital, Lexington, Kentucky
  - Ochsner Clinic Foundation, New Orleans, Louisiana
  - MD Anderson Cancer Center at Cooper, Camden, New Jersey
  - University of New Mexico Cancer Center, Albuquerque, New Mexico
  - Northwell Health Monter Cancer Center, Lake Success, New York
  - Laura and Isaac Perlmutter Cancer Center at NYU Langone, New York, New York
  - SUNY Upstate Medical University, Syracuse, New York
  - Albert Einstein College of Medicine, The Bronx, New York
  - Levine Cancer Institute, Charlotte, North Carolina
  - FirstHealth Outpatient Cancer Center, Pinehurst, North Carolina
  - MetroHealth Medical Center, Cleveland, Ohio
  - The Ohio State University Wexner Medical Center, Columbus, Ohio
  - Columbus NCORP, Columbus, Ohio
  - Stephenson Cancer Center, Oklahoma City, Oklahoma
  - Oklahoma Cancer Specialists and Research Institute, LLC, Tulsa, Oklahoma
  - Willamette Valley Cancer Institute, Eugene, Oregon
  - Northwest Cancer Specialists, P.C., Portland, Oregon
  - Penn Medicine - Jordan Center for Gynecologic Cancer, Philadelphia, Pennsylvania
  - WellSpan Gynecologic Oncology, York, Pennsylvania
  - Women & Infants Hospital of Rhode Island, Providence, Rhode Island
  - Texas Oncology Surgical Specialists - Austin Central, Austin, Texas
  - Texas Oncology - Bedford, Bedford, Texas
  - Texas Oncology - Dallas - Presbyterian Cancer Center, Dallas, Texas
  - The University of Texas Southwestern Medical Center, Dallas, Texas
  - Texas Oncology - Fort Worth Cancer Center, Fort Worth, Texas
  - Texas Oncology - San Antonio Medical Center, San Antonio, Texas
  - Texas Oncology - The Woodlands, The Woodlands, Texas
  - Texas Oncology, Tyler, Texas
- Brazil (12):
  - CRIO - Centro Regional Integrado de Oncologia, Fortaleza, Ceará
  - Hospital Santa Rita, Vitória, Espírito Santo
  - IMIP - Instituto de Medicina Integral Prof. Fernando Figueira, Recife, Pernambuco
  - ONCOSITE/Hospital de Caridade de Ijuí, Ijuí, Rio Grande do Sul
  - Hospital Mãe de Deus, Porto Alegre, Rio Grande do Sul
  - CECOR - Centro Oncológico de Roraima, Boa Vista, Roraima
  - Hospital de CÃ¢ncer de Barretos, Barretos, São Paulo
  - INCA - Instituto Nacional de Câncer, Rio de Janeiro
  - Instituto do Câncer do Estado de São Paulo, São Paulo
  - Perola Centro de Pesquisa em Oncologia, São Paulo
  - Hospital Amaral Carvalho, São Paulo
  - Fundação Antonio Prudente/AC Camargo Cancer Center, São Paulo
- Mexico (4):
  - COI Centro Oncológico Internacional S.A.P.I. de C.V., Mexico City, Mexico City
  - Christus Muguerza Hospital Vidriera, Monterrey, Nuevo León
  - Oaxaca Site Management Organization (OSMO), Oaxaca City
  - Cancerologia De Queretaro, Querétaro
- Clinica MonteSur, Centro de Investigación Clínica Montesur RCI -259, Lima Lima, Peru
- South Korea (3):
  - Seoul National University, Seoul
  - Gangnam Severence Hospital, Seoul
  - Samsung Medical Center, Seoul
- Taiwan (4):
  - Taichung Veterans General Hospital, Taichung
  - Mackay Memorial Hospital Taipei Branch, Taipei
  - Taipei Veterans General Hospital, Taipei
  - Koo Foundation Sun Yat-Sen Cancer Center, Taipei
- Thailand (2):
  - King Chulalongkorn Memorial Hospital, Chulalongkorn University, Bangkok
  - Ramathibodi Hospital, Mahidol University, Bangkok

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Allie SR, Zhang W, Fuse S, Usherwood EJ. Programmed death 1 regulates development of central memory CD8 T cells after acute viral infection. J Immunol. 2011 Jun 1;186(11):6280-6. doi: 10.4049/jimmunol.1003870. Epub 2011 Apr 27. PMID 21525385
- [Result] Antonia S, Goldberg SB, Balmanoukian A, Chaft JE, Sanborn RE, Gupta A, Narwal R, Steele K, Gu Y, Karakunnel JJ, Rizvi NA. Safety and antitumour activity of durvalumab plus tremelimumab in non-small cell lung cancer: a multicentre, phase 1b study. Lancet Oncol. 2016 Mar;17(3):299-308. doi: 10.1016/S1470-2045(15)00544-6. Epub 2016 Feb 6. PMID 26858122
- [Result] Antonia SJ, Lopez-Martin JA, Bendell J, Ott PA, Taylor M, Eder JP, Jager D, Pietanza MC, Le DT, de Braud F, Morse MA, Ascierto PA, Horn L, Amin A, Pillai RN, Evans J, Chau I, Bono P, Atmaca A, Sharma P, Harbison CT, Lin CS, Christensen O, Calvo E. Nivolumab alone and nivolumab plus ipilimumab in recurrent small-cell lung cancer (CheckMate 032): a multicentre, open-label, phase 1/2 trial. Lancet Oncol. 2016 Jul;17(7):883-895. doi: 10.1016/S1470-2045(16)30098-5. Epub 2016 Jun 4. PMID 27269741
- [Result] Barber DL, Wherry EJ, Masopust D, Zhu B, Allison JP, Sharpe AH, Freeman GJ, Ahmed R. Restoring function in exhausted CD8 T cells during chronic viral infection. Nature. 2006 Feb 9;439(7077):682-7. doi: 10.1038/nature04444. Epub 2005 Dec 28. PMID 16382236
- [Result] Borcoman E, Le Tourneau C. Pembrolizumab in cervical cancer: latest evidence and clinical usefulness. Ther Adv Med Oncol. 2017 Jun;9(6):431-439. doi: 10.1177/1758834017708742. Epub 2017 May 8. PMID 28607581
- [Result] Boutros C, Tarhini A, Routier E, Lambotte O, Ladurie FL, Carbonnel F, Izzeddine H, Marabelle A, Champiat S, Berdelou A, Lanoy E, Texier M, Libenciuc C, Eggermont AM, Soria JC, Mateus C, Robert C. Safety profiles of anti-CTLA-4 and anti-PD-1 antibodies alone and in combination. Nat Rev Clin Oncol. 2016 Aug;13(8):473-86. doi: 10.1038/nrclinonc.2016.58. Epub 2016 May 4. PMID 27141885
- [Result] Bristol-Myers Squibb USA, 2017a. Opdivo® (nivolumab) package insert,
- [Result] Bristol-Myers Squibb USA, 2017b. Yervoy® (ipilimumab) package insert,
- [Result] Buchbinder EI, Desai A. CTLA-4 and PD-1 Pathways: Similarities, Differences, and Implications of Their Inhibition. Am J Clin Oncol. 2016 Feb;39(1):98-106. doi: 10.1097/COC.0000000000000239. PMID 26558876
- [Result] Bulliard Y, Jolicoeur R, Windman M, Rue SM, Ettenberg S, Knee DA, Wilson NS, Dranoff G, Brogdon JL. Activating Fc gamma receptors contribute to the antitumor activities of immunoregulatory receptor-targeting antibodies. J Exp Med. 2013 Aug 26;210(9):1685-93. doi: 10.1084/jem.20130573. Epub 2013 Jul 29. PMID 23897982
- [Result] Callahan MK, Wolchok JD, Allison JP. Anti-CTLA-4 antibody therapy: immune monitoring during clinical development of a novel immunotherapy. Semin Oncol. 2010 Oct;37(5):473-84. doi: 10.1053/j.seminoncol.2010.09.001. PMID 21074063
- [Result] Camacho LH. CTLA-4 blockade with ipilimumab: biology, safety, efficacy, and future considerations. Cancer Med. 2015 May;4(5):661-72. doi: 10.1002/cam4.371. Epub 2015 Jan 25. PMID 25619164
- [Result] Carbone DP, Reck M, Paz-Ares L, Creelan B, Horn L, Steins M, Felip E, van den Heuvel MM, Ciuleanu TE, Badin F, Ready N, Hiltermann TJN, Nair S, Juergens R, Peters S, Minenza E, Wrangle JM, Rodriguez-Abreu D, Borghaei H, Blumenschein GR Jr, Villaruz LC, Havel L, Krejci J, Corral Jaime J, Chang H, Geese WJ, Bhagavatheeswaran P, Chen AC, Socinski MA; CheckMate 026 Investigators. First-Line Nivolumab in Stage IV or Recurrent Non-Small-Cell Lung Cancer. N Engl J Med. 2017 Jun 22;376(25):2415-2426. doi: 10.1056/NEJMoa1613493. PMID 28636851
- [Result] Carlino, M.S. et al., 2017. KEYNOTE-029: Efficacy and safety of pembrolizumab (pembro) plus ipilimumab (ipi) for advanced melanoma. In ASCO Annual Meeting. Chicago.
- [Result] Chand D, Savistky D, Gonzalez A,, et al. [Abstract]. J Immunother Cancer. 2017;5(Suppl2):P312.
- [Result] Chemnitz JM, Parry RV, Nichols KE, June CH, Riley JL. SHP-1 and SHP-2 associate with immunoreceptor tyrosine-based switch motif of programmed death 1 upon primary human T cell stimulation, but only receptor ligation prevents T cell activation. J Immunol. 2004 Jul 15;173(2):945-54. doi: 10.4049/jimmunol.173.2.945. PMID 15240681
- [Result] Chung CH. Managing premedications and the risk for reactions to infusional monoclonal antibody therapy. Oncologist. 2008 Jun;13(6):725-32. doi: 10.1634/theoncologist.2008-0012. PMID 18586928
- [Result] Chung HC, Schellens JHM, Delord JP, et al. 2018. Pembrolizumab treatment of advanced cervical cancer: Updated results from the phase 2 KEYNOTE-158 study. [ASCO abstract 5522]. J Clin Oncol. 36(15 suppl):5522.
- [Result] Das R, Verma R, Sznol M, Boddupalli CS, Gettinger SN, Kluger H, Callahan M, Wolchok JD, Halaban R, Dhodapkar MV, Dhodapkar KM. Combination therapy with anti-CTLA-4 and anti-PD-1 leads to distinct immunologic changes in vivo. J Immunol. 2015 Feb 1;194(3):950-9. doi: 10.4049/jimmunol.1401686. Epub 2014 Dec 24. PMID 25539810
- [Result] Disis ML. Immune regulation of cancer. J Clin Oncol. 2010 Oct 10;28(29):4531-8. doi: 10.1200/JCO.2009.27.2146. Epub 2010 Jun 1. PMID 20516428
- [Result] Drescher, C., Moore, M.N., Liu, J., O'Malley, D.M., Wang, E.W., Wang, J.S-Z., Subbish, V., et al. Phase 1/2, Open-Label, Multiple Ascending Dose Trial of AGEN2034, an Anti-PD-1 Monoclonal Antibody, in Advanced Solid Malignancies: Results of Dose Escalation in Advanced Cancer and Expansion Cohorts in Subjects With Relapsed/Refractory Cervical Cancer. Poster presented at European Society for Medical Oncology. Poster presented at ESMO 2018 Congress; 19 - 23 Oct 2018; Munich, Germany; Poster 1158P. Ann Oncol 2018 Oct; 29(Suppl 8).
- [Result] Eggermont AM, Chiarion-Sileni V, Grob JJ, Dummer R, Wolchok JD, Schmidt H, Hamid O, Robert C, Ascierto PA, Richards JM, Lebbe C, Ferraresi V, Smylie M, Weber JS, Maio M, Bastholt L, Mortier L, Thomas L, Tahir S, Hauschild A, Hassel JC, Hodi FS, Taitt C, de Pril V, de Schaetzen G, Suciu S, Testori A. Prolonged Survival in Stage III Melanoma with Ipilimumab Adjuvant Therapy. N Engl J Med. 2016 Nov 10;375(19):1845-1855. doi: 10.1056/NEJMoa1611299. Epub 2016 Oct 7. PMID 27717298
- [Result] Eisenhauer EA, Therasse P, Bogaerts J, Schwartz LH, Sargent D, Ford R, Dancey J, Arbuck S, Gwyther S, Mooney M, Rubinstein L, Shankar L, Dodd L, Kaplan R, Lacombe D, Verweij J. New response evaluation criteria in solid tumours: revised RECIST guideline (version 1.1). Eur J Cancer. 2009 Jan;45(2):228-47. doi: 10.1016/j.ejca.2008.10.026. PMID 19097774
- [Result] Food and Drug Administration. 2018. FDA approves pembrolizumab for advanced cervical cancer with disease progression during or after chemotherapy. https://www.fda.gov/drugs/informationondrugs/approveddrugs/ucm610572.htm. Accessed 14 January 2019.
- [Result] Frenel, J.-S. et al., 2017. Pembrolizumab in patients with advanced cervical squamous cell cancer: Preliminary results from the phase Ib KEYNOTE-028 study. Journal of Clinical Oncology, 34(suppl; abstr 5515).
- [Result] Goldman, J.W. et al., 2017. Nivolumab (N) plus ipilimumab (I) as first-line (1L) treatment for advanced (adv) NSCLC: 2-yr OS and long-term outcomes from CheckMate 012. In ASCO Annual Meeting. Chicago.
- [Result] Gombos RB, Gonzalez A, Manrique M, Chand D, Savitsky D, Morin B, Breous-Nystrom E, Dupont C, Ward RA, Mundt C, Duckless B, Tang H, Findeis MA, Schuster A, Waight JD, Underwood D, Clarke C, Ritter G, Merghoub T, Schaer D, Wolchok JD, van Dijk M, Buell JS, Cuillerot JM, Stein R, Drouin EE, Wilson NS. Toxicological and pharmacological assessment of AGEN1884, a novel human IgG1 anti-CTLA-4 antibody. PLoS One. 2018 Apr 4;13(4):e0191926. doi: 10.1371/journal.pone.0191926. eCollection 2018. PMID 29617360
- [Result] Goodman AM, Kato S, Bazhenova L, Patel SP, Frampton GM, Miller V, Stephens PJ, Daniels GA, Kurzrock R. Tumor Mutational Burden as an Independent Predictor of Response to Immunotherapy in Diverse Cancers. Mol Cancer Ther. 2017 Nov;16(11):2598-2608. doi: 10.1158/1535-7163.MCT-17-0386. Epub 2017 Aug 23. PMID 28835386
- [Result] Hammers HJ, Plimack ER, Infante JR, Rini BI, McDermott DF, Lewis LD, Voss MH, Sharma P, Pal SK, Razak ARA, Kollmannsberger C, Heng DYC, Spratlin J, McHenry MB, Amin A. Safety and Efficacy of Nivolumab in Combination With Ipilimumab in Metastatic Renal Cell Carcinoma: The CheckMate 016 Study. J Clin Oncol. 2017 Dec 1;35(34):3851-3858. doi: 10.1200/JCO.2016.72.1985. Epub 2017 Jul 5. PMID 28678668
- [Result] Hellmann, M.D. et al., 2016. CheckMate 012: safety and efficacy of first-line nivolumab and ipilimumab in advanced NSCLC. In ASCO Annual Meeting. Chicago: Proc Am Soc Clin Oncol.
- [Result] Hellmann MD, Rizvi NA, Goldman JW, Gettinger SN, Borghaei H, Brahmer JR, Ready NE, Gerber DE, Chow LQ, Juergens RA, Shepherd FA, Laurie SA, Geese WJ, Agrawal S, Young TC, Li X, Antonia SJ. Nivolumab plus ipilimumab as first-line treatment for advanced non-small-cell lung cancer (CheckMate 012): results of an open-label, phase 1, multicohort study. Lancet Oncol. 2017 Jan;18(1):31-41. doi: 10.1016/S1470-2045(16)30624-6. Epub 2016 Dec 5. PMID 27932067
- [Result] Hellmann MD, Callahan MK, Awad MM, Calvo E, Ascierto PA, Atmaca A, Rizvi NA, Hirsch FR, Selvaggi G, Szustakowski JD, Sasson A, Golhar R, Vitazka P, Chang H, Geese WJ, Antonia SJ. Tumor Mutational Burden and Efficacy of Nivolumab Monotherapy and in Combination with Ipilimumab in Small-Cell Lung Cancer. Cancer Cell. 2018 May 14;33(5):853-861.e4. doi: 10.1016/j.ccell.2018.04.001. Epub 2018 May 3. PMID 29731394
- [Result] Hellmann MD, Nathanson T, Rizvi H, Creelan BC, Sanchez-Vega F, Ahuja A, Ni A, Novik JB, Mangarin LMB, Abu-Akeel M, Liu C, Sauter JL, Rekhtman N, Chang E, Callahan MK, Chaft JE, Voss MH, Tenet M, Li XM, Covello K, Renninger A, Vitazka P, Geese WJ, Borghaei H, Rudin CM, Antonia SJ, Swanton C, Hammerbacher J, Merghoub T, McGranahan N, Snyder A, Wolchok JD. Genomic Features of Response to Combination Immunotherapy in Patients with Advanced Non-Small-Cell Lung Cancer. Cancer Cell. 2018 May 14;33(5):843-852.e4. doi: 10.1016/j.ccell.2018.03.018. Epub 2018 Apr 12. PMID 29657128
- [Result] Hollebecque, A. et al., 2017. An open-label, multicohort, phase I/II study of nivolumab in patients with virus-associated tumors (CheckMate 358): Efficacy and safety in recurrent or metastatic (R/M) cervical, vaginal, and vulvar cancers. Journal of Clinical Oncology, 35(suppl;abstr 5504).
- [Result] Huang G, Sun X, Liu D, Zhang Y, Zhang B, Xiao G, Li X, Gao X, Hu C, Wang M, Ren H, Qin S. The efficacy and safety of anti-PD-1/PD-L1 antibody therapy versus docetaxel for pretreated advanced NSCLC: a meta-analysis. Oncotarget. 2017 Dec 15;9(3):4239-4248. doi: 10.18632/oncotarget.23279. eCollection 2018 Jan 9. PMID 29423118
- [Result] Jia M, Feng W, Kang S, Zhang Y, Shen J, He J, Jiang L, Wang W, Guo Z, Peng G, Chen G, He J, Liang W. Evaluation of the efficacy and safety of anti-PD-1 and anti-PD-L1 antibody in the treatment of non-small cell lung cancer (NSCLC): a meta-analysis. J Thorac Dis. 2015 Mar;7(3):455-61. doi: 10.3978/j.issn.2072-1439.2015.02.06. PMID 25922725
- [Result] Keytruda [package insert]. Whitehouse Station, NJ; Merck and Co, Inc; 2018.
- [Result] Kumar V, Chaudhary N, Garg M, Floudas CS, Soni P, Chandra AB. Current Diagnosis and Management of Immune Related Adverse Events (irAEs) Induced by Immune Checkpoint Inhibitor Therapy. Front Pharmacol. 2017 Feb 8;8:49. doi: 10.3389/fphar.2017.00049. eCollection 2017. PMID 28228726
- [Result] Larkin J, Hodi FS, Wolchok JD. Combined Nivolumab and Ipilimumab or Monotherapy in Untreated Melanoma. N Engl J Med. 2015 Sep 24;373(13):1270-1. doi: 10.1056/NEJMc1509660. No abstract available. PMID 26398076
- [Result] Latchman Y, Wood CR, Chernova T, Chaudhary D, Borde M, Chernova I, Iwai Y, Long AJ, Brown JA, Nunes R, Greenfield EA, Bourque K, Boussiotis VA, Carter LL, Carreno BM, Malenkovich N, Nishimura H, Okazaki T, Honjo T, Sharpe AH, Freeman GJ. PD-L2 is a second ligand for PD-1 and inhibits T cell activation. Nat Immunol. 2001 Mar;2(3):261-8. doi: 10.1038/85330. PMID 11224527
- [Result] Long, G.V. et al., 2016. Pembrolizumab (pembro) plus ipilimumab (ipi) for advanced melanoma: Results of the KEYNOTE-029 expansion cohort. Journal of Clinical Oncology, 34(15_suppl), pp.9506-9506.
- [Result] Marabelle A, Kohrt H, Sagiv-Barfi I, Ajami B, Axtell RC, Zhou G, Rajapaksa R, Green MR, Torchia J, Brody J, Luong R, Rosenblum MD, Steinman L, Levitsky HI, Tse V, Levy R. Depleting tumor-specific Tregs at a single site eradicates disseminated tumors. J Clin Invest. 2013 Jun;123(6):2447-63. doi: 10.1172/JCI64859. PMID 23728179
- [Result] Mezache L, Paniccia B, Nyinawabera A, Nuovo GJ. Enhanced expression of PD L1 in cervical intraepithelial neoplasia and cervical cancers. Mod Pathol. 2015 Dec;28(12):1594-602. doi: 10.1038/modpathol.2015.108. Epub 2015 Sep 25. PMID 26403783
- [Result] Koh WJ, Greer BE, Abu-Rustum NR, Campos SM, Cho KR, Chon HS, Chu C, Cohn D, Crispens MA, Dizon DS, Dorigo O, Eifel PJ, Fisher CM, Frederick P, Gaffney DK, Han E, Higgins S, Huh WK, Lurain JR 3rd, Mariani A, Mutch D, Nagel C, Nekhlyudov L, Fader AN, Remmenga SW, Reynolds RK, Tillmanns T, Ueda S, Valea FA, Wyse E, Yashar CM, McMillian N, Scavone J. Vulvar Cancer, Version 1.2017, NCCN Clinical Practice Guidelines in Oncology. J Natl Compr Canc Netw. 2017 Jan;15(1):92-120. doi: 10.6004/jnccn.2017.0008. PMID 28040721
- [Result] Oken MM, Creech RH, Tormey DC, Horton J, Davis TE, McFadden ET, Carbone PP. Toxicity and response criteria of the Eastern Cooperative Oncology Group. Am J Clin Oncol. 1982 Dec;5(6):649-55. No abstract available. PMID 7165009
- [Derived] O'Malley DM, Randall LM, Jackson CG, Coleman RL, Hays JL, Moore KN, Naumann RW, Rocconi RP, Slomovitz BM, Tewari KS, Ancukiewicz M, Feliu WO, Monk BJ. RaPiDS (GOG-3028): randomized Phase II study of balstilimab alone or in combination with zalifrelimab in cervical cancer. Future Oncol. 2021 Sep;17(26):3433-3443. doi: 10.2217/fon-2021-0529. Epub 2021 Aug 19. PMID 34409858